CLINICAL TRIAL: NCT04025957
Title: A Phase I Study on Tolerance, Safety and Pharmacokinetics of SHR-1501 in Patients With Advanced Malignancies.
Brief Title: A Study of SHR-1501 in Patients With Advanced Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1501-I-102
Record Dates: First submitted 2019-07-14; First posted 2019-07-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2020-07

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1501 dose escalation (Experimental): SHR-1501 given subcutaneously
  Interventions: Drug: SHR-1501
- SHR-1501 dose expansion (Experimental): SHR-1501 given subcutaneously
  Interventions: Drug: SHR-1501

INTERVENTIONS:
Drug: SHR-1501 — Administered subcutaneously

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of SHR-1501 in patients with advanced malignancies .

ELIGIBILITY:
Inclusion Criteria:

* All Patients All patients must meet all the following criteria to be eligible to participate:

  1. Voluntarily participate in this clinical study, understand the research procedure and be able to sign informed consent in writing;
  2. Subjects must be willing and able to follow the research protocol;
  3. Aged 18-70 years old when the informed consent form is signed;
  4. Have a histologically or cytologically confirmed diagnosis of advanced or metastatic tumor malignancy;
  5. Patients' malignancies must be relapsed or refractory to standard treatment, or patients cannot tolerate standard treatment, or patients have actively refused standard therapy;
  6. Eastern Cooperative Oncology Group ECOG PS score of 0-1;
  7. Have a life expectancy of ≥ 12 weeks;
  8. Adequate organ function defined according to the protocol, These results should be completed within 14 days prior to the first study treatment:
  9. Non-surgically sterilized women of childbearing age or male subjects are required to consent to the use of at least one medically approved contraceptive (eg intrauterine devices, contraceptives or condoms) is performed during the study treatment period and within 3 months of the end of the study treatment period.

Exclusion Criteria:

1. Patients with cancerous meningitis (ie meningeal metastasis);
2. Patients with active central nervous system (CNS) metastasis.
3. Spinal cord compression that cannot be radically treated with surgery and/or radiotherapy cannot be enrolled.
4. Patients with double primary cancers;
5. Patients with a history of autoimmune diseases;
6. Significant clinical significance in the history of cardiovascular disease;
7. Arterial/venous thrombosis events such as cerebrovascular accidents deep vein thrombosis and pulmonary embolism within 6 months prior to first administration;
8. Have a history of immunodeficiency including HIV infection;
9. Active hepatitis B or hepatitis C patients;
10. Any disease or symptom that is not appropriate for inclusion in this study determined by the investigator.;
11. Patients have undergone major surgery within 28 days prior to the first dose (except for diagnostics);
12. Those who used a live attenuated vaccine within 4 weeks prior to the first dose or expect a live attenuated vaccine during the study period;
13. Those who received other clinical trials within 4 weeks prior to the first study;
14. Those who received systemic immunosuppressive therapy within 2 weeks prior to the first study dose;
15. Patients who have previously received allogeneic bone marrow transplantation or solid organ transplantation;
16. A history of severe allergic reactions to other monoclonal antibody/fusion protein drugs;
17. Mental illness, alcohol abuse, drug abuse or substance abuse;
18. Any disease or condition that causes reasonable suspicion to prohibit the use of the study drug or affect the interpretation of the study results or the patient is at high risk of treatment complications (any other disease, metabolic disorder, physical examination results or laboratory tests abnormalities);
19. Pregnant or lactating women or women planning to become pregnant during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Approximately 2 years
  Dose-limiting toxicity in patients with advanced tumors treated by SHR-1501.
Maximum tolerated dose | Approximately 2 years
  Maximum tolerated dose in patients with advanced tumors treated by SHR-1501.
Adverse event/Serious adverse event | Approximately 2 years
  Incidence/severity of adverse events/serious adverse events (rated based on CTC AE v5.0)

SECONDARY OUTCOMES:
Pharmacokinetic (PK) | Approximately 2 years
  Single dose: maximum concentration (Cmax)
Pharmacokinetic (PK) | Approximately 2 years
  Single dose: time to maximum concentration (Tmax)
Pharmacokinetic (PK) | Approximately 2 years
  Single dose: areas under the concentration-time curve (AUClast and AUCinf)
Pharmacokinetic (PK) | Approximately 2 years
  Single dose: half-life (t1/2)
Pharmacokinetic (PK) | Approximately 2 years
  Single dose: clearance (CL)
Pharmacokinetic (PK) | Approximately 2 years
  Single dose: mean residence time (MRT)
Pharmacokinetic (PK) | Approximately 2 years
  Single dose: volume at steady state (Vss)
Pharmacokinetic (PK) | Approximately 2 years
  Multiple doses (at steady state, if applicable): maximum concentration at steady state （Css_max）
Pharmacokinetic (PK) | Approximately 2 years
  Multiple doses (at steady state, if applicable):time to maximum concentration （Tmax）
Pharmacokinetic (PK) | Approximately 2 years
  Multiple doses (at steady state, if applicable):area under the concentration-time curve at steady state （AUCss）
Pharmacokinetic (PK) | Approximately 2 years
  Multiple doses (at steady state, if applicable): t1/2
Pharmacokinetic (PK) | Approximately 2 years
  Multiple doses (at steady state, if applicable):steady-state minimum concentration at steady state （Css_min）
Pharmacokinetic (PK) | Approximately 2 years
  Multiple doses (at steady state, if applicable):average concentration at steady state（Cavg）
Pharmacokinetic (PK) | Approximately 2 years
  Multiple doses (at steady state, if applicable):accumulation ratio （Rac）
Immune-related biomarkers | Approximately 2 years
  indicated by the count of CD8+ T-lymphocytes in peripheral blood at scheduled post-dose time points.
Immune-related biomarkers | Approximately 2 years
  indicated by the percentage of CD8+ T-lymphocytes in peripheral blood at scheduled post-dose time points.
Immune-related biomarkers | Approximately 2 years
  indicated by the count of natural killer (NK) cells in peripheral blood at scheduled post-dose time points.
Immune-related biomarkers | Approximately 2 years
  indicated by the percentage of natural killer (NK) cells in peripheral blood at scheduled post-dose time points.
Objective response rate | Approximately 2 years
  Percentage of participants with CR or PR.
Disease control rate | Approximately 2 years
  Percentage of participants with CR or PR or SD.
Immunogenicity | Approximately 2 years
  The immunogenicity of SHR-1501 single drug. The indicator includes number of participants with anti-drug antibody positive or neutralizing antibody positive.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, MD, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer hospital, Chinese academy of medical sciences, Beijing, China